CLINICAL TRIAL: NCT00304811
Title: Vancomycin Versus Vancomycin Plus Gentamycin For Treating Bacteremic Infection Due to Methicillin-Resistant Staphylococcus Aureus (MRSA)
Brief Title: Vancomycin vs. Vancomycin Plus Gentamycin in Treatment of MRSA Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Collaborators: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: H-17556
Record Dates: First submitted 2006-03-16; First posted 2006-03-20 (Estimated); Last update posted 2009-09-28 (Estimated); Status verified 2009-09

CONDITIONS: Staphylococcus Aureus
Keywords: MRSA; Methicillin Resistant Staphylococcus aureus
MeSH Terms: conditions — Staphylococcal Infections | interventions — Vancomycin; Gentamicins; Rifampin

INTERVENTIONS:
Drug: Vancomycin
Drug: Vancomycin plus Gentamicin
Drug: Vancomycin plus Rifampin
Drug: Vancomycin plus Gentamicin plus Rifampin

SUMMARY:
The purpose of this study is to compare the outcome of treatment for bacteremic MRSA infection with vancomycin alone, vancomycin plus gentamicin, vancomycin plus rifampin, and vancomycin plus gentamicin and rifampin.

DETAILED DESCRIPTION:
Treatment of bacteremic infection (infection associated with positive blood cultures) due to Staphylococcus aureus has become increasingly problematic as a result of the increasing prevalence of strains that are resistant to beta-lactam antibiotics (so-called methicillin-resistant Staphylococcus aureus, MRSA). About 70% of hospital-related strains of S. aureus are MRSA, and, in the past 4 years, the incidence of MRSA in community-acquired infection has risen to about 50%; these data are quite representative of what is being seen elsewhere in the United States and other parts of the world.

Bacteremic MRSA infections are highly problematic for at least two reasons: (1)they are serious, with substantial morbidity and about a 25% rate of mortality in middle-aged adults, the principal patients in our system; and (2)available antibiotic therapy is suboptimal.

In the pre-MRSA era (before 1982 in the United States), treatment of bacteremic S. aureus infection with a beta-lactam antibiotic such as nafcillin produced a uniform microbiological cure (Musher DM, McKenzie SO: Infections due to Staphylococcus aureus. Medicine 56:383-409, 1977). This means that, in the absence of an untreated focus of infection that required surgical removal (such as a myocardial abscess), antibiotics rapidly sterilized the blood stream. This does not mean that no one died; deaths from complications of infection remained common. But, at autopsy, there was generally no evidence for active infection. Extensive literature examined the question of whether gentamicin should be added to nafcillin to treat this kind of disease (reviewed critically in DM, Verner EF: Treatment of Infections due to Staphylococcus aureus. IN The Staphylococci, Ed. by J Jeljascewicz, Gustave Fischer Verlag, Stuttgart, New York, pp.407-419, 1986). Gentamicin produced a synergistic bactericidal effect agains S. aureus in vitro and in animal models. In humans, the addition of gentamicin was associated with more rapid sterilization of the blood stream, but prolonged gentamicin therapy was also associated with nephrotoxicity.

In contrast, in the MRSA era, treatment with vancomycin is associated with persistence of bacteremia (positive blood cultures) and death from active infection. We have recently participated in a prospective observational study that documented the association between vancomycin treatment, persistently positive blood cultures, and persistence of active infection during treatment of S. aureus bacteremia with vancomycin (Chang F-Y, McDonald BB, Peacock, Jr. JE, Musher DM, et al. Staphylococcus aureus bacteremia: recurrence and the impact of antibiotic treatment in a prospective multicenter study. Medicine 82:333-339, 2003).

There appears to be a very close correlation between the outcome of treatment for serious S. aureus infection and the bactericidal activity of the treating antibiotic in vitro using conventional techniques (Musher DM, Verner EF: Treatment of infections due to Staphylococcus aureus. IN The Staphylococci, Ed. by J Jeljascewicz, Gustave Fischer Verlag, Stuttgart, New York, pp.407-419, 1986). We recently showed that adding low concentrations of gentamicin to vancomycin led to substantial synergistic bactericidal activity against MRSA (Shelburne SA, Musher DM, Hulten K, Ceasar H, Lu MY, Bhaila I, Hamill RJ. In-vitro killing of community-associated methicillin-resistant Staphylococcus aureus with drug combinations. Antimicrob Agents Chemother 48:4016-9, 2004).

Based in part on the analogy of nafcillin for treating methicillin-susceptible S. aureus infection, and in part of in vitro studies such as ours (cited above), some physicians regularly add gentamicin to vancomycin for treating MRSA infection. Others, without even the in vitro support, add rifampin either instead of gentamicin or together with gentamicin. There are no clinical studies to support or to refute any of these clinically motivated usages.

Thus, at present, about one-third of patients with MRSA bacteremia at VAMC are treated with vacomycin plus gentamicin, and two-thirds receive vancomycin alone; some in each group receive rifampin. The decisionto add gentamicin is made a haphazard fashion. Our proposal is, once MRSA has been identified in acceptable regimens by stratifying patients prospectively to vancomycin alone or vancomycin plus gentamicin, and further stratifying each of those groups to be with or without rifampin.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MRSA in a blood culture processed as standard of care at the VAMC
* Patients or next of kin willing to sign consent to be randomized by social security number to one of the treatments.

Exclusion Criteria:

* none

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2006-01; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Time to defervescence (24 hours of temperature <100 degrees F)
Return of WBC to normal (<10,500)
negative blood cultures
discharge

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Musher, MD, Principal Investigator — Baylor College of Medicine, Houston VA Medical Center
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas